CLINICAL TRIAL: NCT05980507
Title: An Open Label, Single-arm Clinical Study Evaluating the Safety and Efficacy of ICI201 Infusion in Relapsed/Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Molecular development strategy adjustment
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICI201Y001
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICI201 (Experimental)
  Interventions: Drug: ICI201

INTERVENTIONS:
Drug: ICI201 — ICI201 CAR-T cell injection

SUMMARY:
An open label, single-arm clinical study evaluating the safety and efficacy of ICI201 infusion in relapsed/refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* 1. According to the multiple myeloma diagnostic criteria of the International Myeloma Working Group (IMWG), there is the initial diagnosis of multiple myeloma. 2. Subjects must have previously received at least 3 anti-myeloma regimens. Subjects must have documented disease progression (according to IMWG criteria) during or within 12 months of completing their last anti-myeloma regimen prior to study entry; and prior regimens must have included proteasome inhibitor (PI) and immunomodulatory drug (IMiD). 3. Measurable disease as defined by the protocol 4. ECOG score is 0 or 1. 5. Expected survival time ≥12 weeks. 6. GPRC5D positive expression in bone marrow plasma cells

Exclusion Criteria:

* 1. Patients suffering from graft-versus-host disease (GVHD) or requiring immunosuppressants drugs. 2. Patients who received autologous hematopoietic stem cell transplantation (ASCT) or prior allogeneic hematopoietic stem cell transplantation (ALLo-HSCT) within 12 weeks prior to mononuclear cell collection. 3. Screening subjects who were receiving systemic steroids during the previous 7 days or who were determined by the investigator to require long-term systemic steroid use during treatment (except for inhaled or topical use, except at doses < 10mg/ day). 4. Patients with a history of hypertension that cannot be controlled by medication (blood pressure ≥140/90 mmHg). 5. Patients who have recieved GPRC5D-targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-18 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Time Frame: 28 days post ICI201 administration
  Dose limiting toxicity (DLT)
Incidence and severity of all adverse events related to study drug | Time Frame: 2 years post ICI201 administration
  Incidence and severity of all adverse events related to study drug

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China